CLINICAL TRIAL: NCT02698163
Title: Nanodiamond Modified Gutta Percha (NDGP) Composite for Non-surgical Root Canal Therapy (RCT) Filler Material Applied by Vertical Condensation Obturation Procedure
Brief Title: Nanodiamond Modified Gutta Percha (NDGP) Composite for Non-surgical Root Canal Therapy (RCT) Filler Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Eric Sung, DDS, Professor of Clinical Dentistry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-002015
Record Dates: First submitted 2016-02-25; First posted 2016-03-03 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Dental Pulp Diseases; Dental Pulp Necrosis; Nerve Root Pain Nec
Keywords: Root Canal Therapy
MeSH Terms: conditions — Dental Pulp Diseases; Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gutta Percha (Active Comparator): For all the patients in the control arm of the study, standard treatment of care procedures will be given. Root canal therapy will be given according to the vertical obturation technique. The root canals will be filled with standard root canal filler material: gutta percha at the apical third up to and including the coronal third. The tooth will be restored with a crown for posterior teeth, or a composite filling for anterior teeth.
  Interventions: Device: Gutta Percha
- Nanodiamond reinforced Gutta Percha (Experimental): For all the patients in the treatment arm of the study, standard treatment of care procedures will be given. Root canal therapy will be given according to the vertical obturation technique. The difference between the two arms will be the root canal filler material used. The root canals for the treatment arm of the study will be filled with gutta percha at the apical third, Nanodiamond gutta percha (NDGP) in the middle third, and again with gutta percha at the coronal third. The tooth will be restored with a crown for posterior teeth, or a composite filling for anterior teeth.
  Interventions: Device: Nanodiamond reinforced Gutta Percha; Device: Gutta Percha

INTERVENTIONS:
Device: Nanodiamond reinforced Gutta Percha — Gutta percha reinforced with 5 nm diameter nanodiamonds 5 wt % (NDGP).
  Other Names: NDGP
  Arms: Nanodiamond reinforced Gutta Percha
Device: Gutta Percha — Gutta percha is a device made from coagulated sap of certain tropical trees intended to fill the root canal of a tooth. The gutta percha is softened by heat and inserted into the root canal, where it hardens as it cools. Gutta percha is classified as Class I (general controls).
  Other Names: GP

SUMMARY:
Non-surgical root canal therapy (RCT) represents a standard of treatment that addresses infected pulp tissue in teeth and protects against future infection while preserving the tooth for the patient for mainly cosmetic purposes. RCT is offered as the better cosmetic, cheaper, and less time intensive treatment option for a patient compared to those of dental implantation. Dental implantation is the alternative to RCT, and they are both originally offered at the time of the initial consultation. RCT involves non-surgically removing dental pulp comprising blood vessels and nerve tissue, decontaminating residually infected tissue, and using a filler material to replace the non-surgically created space where the pulp was removed. Currently, standard of care treatment for RCT utilizes gutta-percha as the root canal filling material. Our research group has previously demonstrated NDGP's improvement in tensile strength compared to those of gutta-percha. This research studies a new type of filler, gutta-percha modified by the addition of nanodiamond material (NDGP). This is an equivalence study of NDGP and standard gutta-percha administration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older when patient is referred to UCLA endodontics department for root canal therapy
* Patient referral to UCLA endodontics department for root canal therapy

Exclusion Criteria:

* preoperative periodontal disease
* prior non-surgical and surgical endodontic treatment
* currently taking medications used to treat osteoporosis or any form of IV biphosphonates
* allergic to dental materials
* dental phobia
* MD consult/medically compromised/prophylaxis needed
* developmental/congenital disorders
* craniofacial disorder/syndromic cases
* low pain tolerance ascertained from past dental experience
* current moderate to severe periodontitis
* previous RCT/initiated pulp therapy
* previous apical surgery
* previous surgical root canal procedure
* with psychiatric and/or mental health history
* poor oral hygiene
* poor diet
* illicit and/or recreational drug use
* complicated dental history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Ho, M.S., Ph.D., Principal Investigator — University of California, Los Angeles; Mo K Kang, Ph.D.,D.D.S., Principal Investigator — University of California, Los Angeles; Eric C Sung, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee DK, Kim SV, Limansubroto AN, Yen A, Soundia A, Wang CY, Shi W, Hong C, Tetradis S, Kim Y, Park NH, Kang MK, Ho D. Nanodiamond-Gutta Percha Composite Biomaterials for Root Canal Therapy. ACS Nano. 2015 Nov 24;9(11):11490-501. doi: 10.1021/acsnano.5b05718. Epub 2015 Oct 15. PMID 26452304

RESULTS

PARTICIPANT FLOW:
Groups:
- Gutta Percha: For all the patients in the control arm of the study, standard treatment of care procedures will be given. Root canal therapy will be given according to the vertical obturation technique. The root canals will be filled with standard root canal filler material: gutta percha at the apical third up to and including the coronal third. The tooth will be restored with a crown for posterior teeth, or a composite filling for anterior teeth. One tooth per participant was treated.
  Gutta Percha: Gutta percha is a device made from coagulated sap of certain tropical trees intended to fill the root canal of a tooth. The gutta percha is softened by heat and inserted into the root canal, where it hardens as it cools. Gutta percha is classified as Class I (general controls).
- Nanodiamond Reinforced Gutta Percha: For all the patients in the treatment arm of the study, standard treatment of care procedures will be given. Root canal therapy will be given according to the vertical obturation technique. The difference between the two arms will be the root canal filler material used. The root canals for the treatment arm of the study will be filled with gutta percha at the apical third, Nanodiamond gutta percha (NDGP) in the middle third, and again with gutta percha at the coronal third. The tooth will be restored with a crown for posterior teeth, or a composite filling for anterior teeth.
  Nanodiamond reinforced Gutta Percha: Gutta percha reinforced with 5 nm diameter nanodiamonds 5 wt % (NDGP).
  Gutta Percha: Gutta percha is a device made from coagulated sap of certain tropical trees intended to fill the root canal of a tooth. The gutta percha is softened by heat and inserted into the root canal, where it hardens as it cools. Gutta percha is classified as Class I (general controls). One tooth per participant was treated.
Period: Overall Study
Arm/Group | Gutta Percha | Nanodiamond Reinforced Gutta Percha
Started | 1 | 3
Completed | 1 | 2
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gutta Percha | Nanodiamond Reinforced Gutta Percha | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (0) | 67 (21.66) | 68.25 (17.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Apical Radio-lucency
Description: A radiograph of the treated tooth is made after 6 months post treatment, which will be compared with the radiograph of the treated tooth taken immediately after the RCT procedure. Clinical examination is performed at 6 months after the operation. The greatest diameters (mm) of the radio-lucency were recorded.
Time Frame: 6 months
Population: One of the recruited patients in the Nanodiamond reinforced Gutta Percha group failed to follow up.
Measure: Mean (Standard Deviation); unit: % Change in Diameter (mm)
Arm/Group | Gutta Percha | Nanodiamond Reinforced Gutta Percha
Number analyzed (Participants) | 1 | 2
% Change in Diameter (mm) | 17.4 (0) | 27.1 (4.6)

2. Primary Outcome: Number of Participants With Absence of Apical Periodontitis
Description: Apical periodontitis resulting in pain and apical lucency is measured. A radiograph of the treated tooth is made after 1 year post treatment, which will be compared with the radiographs of the treated tooth taken immediately after the RCT procedure and 6 months post treatment. Clinical examination is performed at 1 year after the operation.
Time Frame: 1 year
Population: One of the recruited patients in the Nanodiamond reinforced Gutta Percha group failed to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Gutta Percha | Nanodiamond Reinforced Gutta Percha
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

3. Secondary Outcome: Number of Participants With Post-Operative Pain
Description: Clinical examination is performed at 6 month after the operation to determine post-operative pain. Pain was assessed via a postoperative survey and a clinical examination (comparative pain scale 0 - 10; 0 is no pain and 10 is spontaneous pain).
Time Frame: 6 months
Population: One of the recruited patients in the Nanodiamond reinforced Gutta Percha group failed to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Gutta Percha | Nanodiamond Reinforced Gutta Percha
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Tooth Survival (6 Month)
Description: A radiograph of the treated tooth is made after 6 months post treatment, which will be compared with the radiograph of the treated tooth taken immediately after the RCT procedure. Clinical examination is performed at 6 months after the operation.
Time Frame: 6 months
Population: One of the recruited patients in the Nanodiamond reinforced Gutta Percha group failed to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Gutta Percha | Nanodiamond Reinforced Gutta Percha
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

5. Secondary Outcome: Number of Participants With Tooth Survival (1 Year)
Description: A radiograph of the treated tooth is made after 1 year post treatment, which will be compared with the radiographs of the treated tooth taken immediately after the RCT procedure and 6 months post treatment. Clinical examination is performed at 1 year after the operation.
Time Frame: 1 year
Population: One of the recruited patients in the Nanodiamond reinforced Gutta Percha group failed to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Gutta Percha | Nanodiamond Reinforced Gutta Percha
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at 3-month and 6-month follow-ups.
Arm/Group | Gutta Percha | Nanodiamond Reinforced Gutta Percha
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT02698163/Prot_SAP_000.pdf